CLINICAL TRIAL: NCT00365924
Title: A Pilot Methodology Study To Evaluate Changes In Bone Quality Parameters Following Therapy With Recombinant Human Parathyroid Hormone, PTH (Forteo)
Brief Title: A Pilot Methodology Study To Evaluate Changes In Bone Quality Parameters Following Therapy With Forteo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A9001294
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2008-06

CONDITIONS: Osteoporosis
Keywords: 12 month therapy with postmenopausal women with osteoporosis to examine changes in bone quality parameters
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Forteo (Other)
  Interventions: Drug: Forteo

INTERVENTIONS:
Drug: Forteo — Open label single arm study with Forteo as an intervention
  Other Names: Recombinant Human PTH 1-34

SUMMARY:
This methodology trial will be conducted in patients with osteoporosis and will measure the changes in bone quality parameters, micro- and macroarchitecture, bone biomarkers and bone density following therapy with the approved drug, Forteo.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with osteoporosis

Exclusion Criteria:

* Any therapies or products affecting bone turnover within 12 months of Screening.
* Bisphosphonate treatment >1 month in total duration at any time in the past.
* In addition, patients must be bisphosphonate-treatment-free for at least 12 months prior to Screening.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Changes in bone quality parameters (micro- and macroarchitecture) in osteoporotic postmenopausal women following 12 months of therapy with Forteo | 12 months

SECONDARY OUTCOMES:
Changes in BMD and bone biomarkers following 12 months of therapy with Forteo | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Argentina (2):
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Capital Federal - Buenos Aires

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001294&StudyName=A%20Pilot%20Methodology%20Study%20To%20Evaluate%20Changes%20In%20Bone%20Quality%20Parameters%20Following%20Therapy%20With%20Forteo